CLINICAL TRIAL: NCT00155402
Title: Phase 1 Study of Applying Fibrin Glue in Patients With Corneal Ulcer or Patients Requiring Wound Closure by Suture
Brief Title: The Application of Fibrin Glue in Ocular Surface Diseases
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Short of supply of fibrin glue
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wei-Li Chen/Assistant Professor, National Taiwan University, Department of Ophthalmology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 940208
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2005-03

CONDITIONS: Pterygium; Corneal Ulcer
Keywords: fibrin glue; corneal perforation; pterygium; conjunctiva; corneal ulcer
MeSH Terms: conditions — Pterygium; Corneal Ulcer; Corneal Perforation | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Use of fibrin glue after corneal surgery or transplantation
  Interventions: Drug: tissue fibrin glue application (Tisseel)

INTERVENTIONS:
Drug: tissue fibrin glue application (Tisseel) — Apply several droplets within several seconds to several minutes

SUMMARY:
This clinical trial tries to use tissue fibrin glues (Tisseel) to treat various ocular surface diseases or surgeries, which includes pterygium surgery, corneal melting/perforation, Gunderson's flap, conjunctival laceration, and muscle/clinical/filtering surgery.

DETAILED DESCRIPTION:
This clinical trial tries to use tissue fibrin glues (Tisseel) to treat various ocular surface diseases or surgeries. The inclusion criteria are:

1. ocular surface disease which may need amniotic membrane transplantation (corneal pro epithelization, pterygium surgery, etc)
2. infectious or noninfectious corneal ulcer with perforation less than 3 mm
3. conjunctival transplantation/suture
4. corneal surgeries which can be treated by conventional suture technique or application with cyanoacrylic acid tissue glues.

Informed consents will be obtained from the patients before applications. After surgeries, topical steroids and antibiotics will be used, and therapeutic contact lens will be used. The patients will be followed up for at least three months.

ELIGIBILITY:
Inclusion Criteria:

* Ocular surface diseases, which are expected to be treated by tissue fibrin glues

Exclusion Criteria:

* Pregnancy
* Children younger than 3 years old

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-04; Study Completion 2008-03

PRIMARY OUTCOMES:
cure of the diseases | 1week, 2 weeks, 3 weeks, 4 weeks

SECONDARY OUTCOMES:
integrity of the ocular surface | 1week, 2 weeks, 3 weeks, 4 weeks
visual acuity | 1week, 2 weeks, 3 weeks, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fung-Rong Hu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Wei-Li Chen, Dawan, Taiwan